CLINICAL TRIAL: NCT04395573
Title: Real Time 3D Navigation and Traditional US to Identify Epidural Space Depth in Obese Pregnant
Acronym: Accuro
Status: Completed | Type: Observational
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: EESOA6
Record Dates: First submitted 2020-05-14; First posted 2020-05-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy Related; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Accuro — ultrasound device (Accuro, Rivanna Medical, Charlottesville, VA) with automated pattern recognition software programmed (SpineNav3DTM technology) to calculate the depth to epidural space and identify bony landmarks
  Other Names: wireless portable ultrasound device
Device: standard ultrasound device — standard ultrasound device (o calculate the depth to epidural space and identify bony landmarks

SUMMARY:
The aim of this study is to assess the accuracy of the Accuro Ultrasound Device in estimating the epidural space depth compared to the Standard Ultrasound Examination and with the measured needle depth during epidural and spinal insertion in pregnant obese patients

DETAILED DESCRIPTION:
SpineNav3DTM technology facilitates image interpretation of individual 2D lumbar spine scans by automating spinal bone landmark detection and depth measurements and providing a real-time assessment of scan plane orientation in 3D.

All the subjects will have their lumbar area scanned for the measurements of the depth of the epidural space (recorded in cm) by two blinded anesthesiologists, one using standard ultrasounds and the other the Accuro Device.

All measurements will be performed either in the sitting or in the supine position at L1/L2, L2/L3 and L3/L4 levels. Neuraxial anesthesia will be performed by using the previously marked interspace by a blinded anesthesiologist who will measure the epidural space depth during epidural or spinal insertion by marking the needle.

ELIGIBILITY:
Inclusion Criteria:

* ASA Status >III
* obese BMI>30
* term gestatio > 37 weeks
* singleton pregnancy
* undergoing elective cesarean section with spinal anesthesia
* requesting epidural labor analgesia

Exclusion Criteria:

* contraindications to neuraxial block
* severe scoliosis
* previous spine surgery

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant patients
Study Population: Pregnant Patients undergoing elective cesarean section or requesting labor epidural analgesia
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Epidural space depth | up to 30 minutes
  the depth of the epidural space (recorded in cm) is defined as the distance from the skin to the posterior complex

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- ASST S Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seligman KM, Weiniger CF, Carvalho B. The Accuracy of a Handheld Ultrasound Device for Neuraxial Depth and Landmark Assessment: A Prospective Cohort Trial. Anesth Analg. 2018 Jun;126(6):1995-1998. doi: 10.1213/ANE.0000000000002407. PMID 28858898